CLINICAL TRIAL: NCT02333526
Title: Soluble Syndecan 1 as Biomarker for Acute and Chronic Bowel Inflammation
Brief Title: Syndecan 1 as Biomarker for Inflammation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Helios Albert-Schweitzer-Klinik Northeim (Other)
Responsible Party: Principal Investigator, Tobias Meister, Priv.-Doz. Dr. med. Tobias Meister, Helios Albert-Schweitzer-Klinik Northeim
Other Study IDs: Syndecan-NOM
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Colitis
Keywords: ulcerative colitis; Clostidium difficile-associated colitis; Syndecan-1; biomarker
MeSH Terms: conditions — Colitis; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — blood serum for soluble Syndecan 1 and CRP Leucocyte cound Blood panel Stool analysis for calprotectin
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to evaluate the soluble biomarker syndecan-1 (sSdc1) taken from venous blood of patients with infectious intestinal diseases such as Clostridium difficile-associated colitis, bacterial colitis, Norovirus enteritis and Crohn´s disease or ulcerative colitis. The level of sSdc1 will be compared with disease activity in patients with active inflammation and with disease in remission. Secondary objectives were the assessment of correlation of the above-mentioned factors with the CRP value. Subjects will be volunteers. Blood will be taken as part of the routine clinical work-up after the written agreement blood and sSdc1-level will be assessed using a human-specific sSdc1 ELISA assay. In addition, the subjects are asked to answer a short questionnaire. The study is designed as a prospective, comparative cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Subject with at least 18 years of age
* able to give informed consent
* healthy volunteer or inflammatory bowel condition (inflammatory bowel disease, infectious colitis)

Exclusion Criteria:

* not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with inflammatoy bowel disease, infectious colitis and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Soluble serum Syndecan-1 in ng/ml | 6 months

SECONDARY OUTCOMES:
Underlying disease | 6 months
Patient age | 6 Months
Disease activity in Inflammatory bowel disease | 6 Months
Calprotectin in stool | 6 Months
Leucocyte blood count | 6 Months
CRP in serum | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Meister, PD Dr.med., Principal Investigator — Helios Albert-Schweitzer-Klinik Northeim
Locations (2):
- Germany (2):
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - Helios Albert-Schweitzer-Klinik Northeim, Northeim, Lower Saxony

REFERENCES:
- [Derived] Floer M, Clausen M, Meister T, Vollenberg R, Bettenworth D, Tepasse PR. Soluble syndecan-1 as marker of intestinal inflammation: A preliminary study and evaluation of a new panel of biomarkers for non-invasive prediction of active ulcerative colitis. Adv Clin Exp Med. 2021 Jul;30(7):655-660. doi: 10.17219/acem/139040. PMID 34286513